CLINICAL TRIAL: NCT06279312
Title: The Effect of Adaptogen Elixir on Sleep Improvement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: N202311065
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Sleep Disorder; Anxiety Disorders
Keywords: Adaptogen
MeSH Terms: conditions — Sleep Wake Disorders; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo drink (Placebo Comparator): consume 1 drink per day for 4 weeks
  Interventions: Dietary Supplement: Placebo drink
- Adaptogen Elixir drink (Experimental): consume 1 drink per day for 4 weeks
  Interventions: Dietary Supplement: Adaptogen Elixir drink

INTERVENTIONS:
Dietary Supplement: Placebo drink — consume 1 drink per day for 4 weeks
  Arms: Placebo drink
Dietary Supplement: Adaptogen Elixir drink — consume 1 drink per day for 4 weeks
  Other Names: Isagenix-Adaptogen Elixir
  Arms: Adaptogen Elixir drink

SUMMARY:
This study aims to examine the effectiveness of Adaptogen Elixir herbal drink in relieving emotions and improving sleep quality. Participants will be randomly assigned to either the placebo group or the Adaptogen Elixir herbal drink group, with 25 participants in each group. On the day of the experiment (week 0), participants are required to collect blood and saliva samples, fill out questionnaires assessing sleep disorders and stress condition, and use a sleep monitoring system to track their sleep and autonomic nervous system conditions. Subsequently, participants will be given the experimental samples and instructed to consume them continuously for 4 weeks following the instruction. Follow-up assessments will be conducted in the 2nd and 4th weeks, participants are required to collect blood and saliva samples, fill out questionnaires assessing sleep disorders and stress condition, and use a sleep monitoring system to track their sleep and autonomic nervous system conditions.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged above 18 years old.
* Individuals experiencing insomnia issues (PSQI > 5) or high levels of anxiety (GAD-7 > 9).
* No medication use or regular use of sleeping pills or antidepressants in the past month.
* No ongoing mental illnesses.
* No ongoing physical illnesses.
* No other sleep disorders.
* No circadian rhythm issues.
* No consumption of sleep or stress-related supplements in the past month.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Individuals with significant organic diseases such as organ transplants, epilepsy or seizures, liver or kidney diseases, malignant tumors, endocrine disorders, or a history of alcohol or substance use disorders.
* Individuals known to be allergic to any components of the product.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2024-02-26 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Sleep monitoring | Week 0 (Baseline), Week 2, Week 4
  The difference of electrocardiosignal between two specific points on the body surface will be used to reflect sleep state.
Sleeping qualityy | Week 0 (Baseline), Week 2, Week 4
  The Pittsburgh Sleep Quality Index (PSQI) will be utilized to assess sleeping quality. The minimum value is 0, the maximum value is 42. The higher the score, the worse the outcome.
Sleeping disorders | Week 0 (Baseline), Week 2, Week 4
  Insomnia Severity Index (ISI) will be utilized to assess sleeping disorders. The minimum value is 0, the maximum value is 28. The higher the score, the worse the outcome.

SECONDARY OUTCOMES:
Neuropeptide Y concentration | Week 0 (Baseline), Week 2, Week 4
  Venous blood samples will be collected to measure concentrations of Neuropeptide Y.
Cortisol concentration | Week 0 (Baseline), Week 2, Week 4
  Saliva samples will be collected to measure concentrations of cortisol.
Anxiety | Week 0 (Baseline), Week 2, Week 4
  Generalized Anxiety Disorder-7 (GAD-7) will be utilized to assess anxiety. The minimum value is 0, the maximum value is 21. The higher the score, the worse the outcome.
Low Frequency/High Frequence (LF/HF) ratio | Week 0 (Baseline), Week 2, Week 4
  A sleep monitoring system will be utilized to measure LF/HF ratio

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-Chien Lee, Doctor, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No